CLINICAL TRIAL: NCT03187392
Title: Topical Lidocaine-prilocaine Cream Versus Lidocaine Infiltration for Pain Relief During Insertion of Subcutaneous Birth Control Implants : A Randomized Controlled Trial
Brief Title: Pain Relief for Birth Control Implants Insertion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Armia Michael, resident physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123456
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Contraception; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine injection (Active Comparator)
  Interventions: Drug: Lidocaine Injectable Product
- lidocaine-prilocaine cream (Experimental)
  Interventions: Drug: Lidocaine Topical Cream [LMX]

INTERVENTIONS:
Drug: Lidocaine Injectable Product — 3 cm of Lidocaine- will be injected subcutaneous for 5 minutes before insertion of subcutaneous birth control implant
  Arms: lidocaine injection
Drug: Lidocaine Topical Cream [LMX] — 3 mg of Lidocaine- will be applied to skin for 5 minutes before insertion of subcutaneous birth control implant
  Arms: lidocaine-prilocaine cream

SUMMARY:
The aim of our study is to compare the analgesic effect of topical application of lidocaine-prilocaine cream and lidocaine infiltration during insertion of birth control implants

ELIGIBILITY:
Inclusion Criteria:

* female want use subcutaneous birth control

Exclusion Criteria:

* previous scar at side of insertion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-09-16 (Estimated); Study Completion 2018-09-18 (Estimated)

PRIMARY OUTCOMES:
Mean pain score during insertion of implant | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No